CLINICAL TRIAL: NCT01630421
Title: Identification of Mutations That Lead to Aplasia Cutis Congenita in Families and Isolated Cases and Studies of Cellular and Molecular Mechanisms
Brief Title: Genetic and Functional Analysis of Aplasia Cutis Congenital (ACC)
Acronym: ACC
Status: Recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Ernst Reichenberger, Assoc. Prof., UConn Health
Other Study IDs: UCHC03-008ACC
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Aplasia Cutis Congenita
Keywords: Aplasia cutis congenita; bone; osteoblast; osteoclast; skin
MeSH Terms: conditions — Ectodermal Dysplasia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, bone tissue, skin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- affected, unaffected: Individuals with diagnosed ACC

SUMMARY:
The goal of this research study is to identify genes and regulatory elements on chromosomes that cause ACC. The investigators also study tissue samples from patients to learn about the processes that lead to this disorder.

DETAILED DESCRIPTION:
Aplasia cutis congenita (ACC) or congenital scalp defect is a very rare disorder that affects bone and skin. The definition for ACC is the localized absence of (normal) skin at the time of birth (congenital). The skin appears thinner and the underlying structures are visible. We study mostly the isolated form of ACC with the lesion often being at the vertex of the skull (at or close to the top of the skull). The bone underlying the lesion is sometimes thinner as well.

For this study we will:

* Send out study participation kits and consent by phone
* Collect a saliva sample from eligible individuals
* Obtain information regarding ACC
* Document disorder with photos and doctor's letters
* If patients undergo surgery for ACC we ask to obtain some tissue that would otherwise be discarded
* Isolate DNA from the saliva sample
* Perform genetic analyses of the DNA with the most up-to-date methods available to identify genetic variations
* Study in the laboratory why the genetic variations cause the disorder

ELIGIBILITY:
Inclusion Criteria:

* ACC; unaffected individuals only if part of a participating ACC family

Exclusion Criteria:

* No ACC unaffected individuals only as part of a participating ACC family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with diagnosed ACC
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic elements | at time of identification
  The goal is to identify relevant genes or genetic elements that cause the disease or contribute to the disease progression and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst J Reichenberger, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Levine SM, Reformat DD, Thorne CH. Cutis aplasia: perioperative management and case report. Am J Crit Care. 2012 May;21(3):212-5. doi: 10.4037/ajcc2012904. PMID 22549580
- See also: Brief description — http://omim.org/entry/107600
- See also: Reichenberger lab research information — https://health.uconn.edu/reichenberger-lab/